CLINICAL TRIAL: NCT01284322
Title: OPEN LABEL TRIAL OF ANTI-TGF-BETA MAB, FRESOLIMUMAB, IN SYSTEMIC SCLEROSIS - A PHASE ONE BIOMARKER TRIAL
Brief Title: Fresolimumab In Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Robert Lafyatis, MD, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H30142
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Diffuse Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fresolimumab (Experimental)
  Interventions: Drug: Fresolimumab

INTERVENTIONS:
Drug: Fresolimumab — intravenous fresolimumab 1mg/kg, first 8 patients; 5 mg/kg following 8 patients
  Other Names: GC1008; anti-TGF-beta

SUMMARY:
The purpose of this study is to determine if fresolimumab is safe in treating people with systemic sclerosis (scleroderma) and to investigate the effect of fresolimumab in the skin of these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Meet ACR criteria for diffuse systemic sclerosis
* < 24 months since onset of first SSc manifestation other than Raynaud's phenomenon
* Modified Rodnan Skin Score ≥ 15
* Male or female adult ( ≥ 18 years of age)
* Able and willing to give written informed consent and comply with study protocol

Exclusion Criteria:

* Moderate or severe pulmonary disease w/ FVC < 80% or DLCO < 70% or ground glass and fibrosis > 20% of lung fields by HRCT
* Treatment with investigational drug within 4 weeks of screening
* Ongoing use of high dose steroids (> 10mg/day) or unstable steroid dose in past 4 weeks
* Treatment with immunosuppressive, cytotoxic, or antifibrotic drug within 4 weeks of screening
* Positive for HIV, HBV, and/or HCV
* Known active infection (bacterial, viral, fungal, mycobacterial, or other); not including fungal infection of nail beds or any major infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening
* Patients w/ history of malignancy or premalignant lesion
* History of keratoacanthoma or squamous cell carcinoma
* Moderate to severe hepatic impairment
* SSc renal crisis within 6 months or creatinine > 2.0
* Lack of IV access for medication administration
* Moderate or severe cardiac disease with significant arrhythmia, heart failure, or unstable angina
* Anemia (Hb < 8.5 gm/dL)
* Thrombocytopenia or blood clotting disorder
* Patients with organ transplant (including allogeneic bone marrow transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate safety of fresolimumab in patients with scleroderma | 24 weeks
To investigate the effect of fresolimumab on TGF-beta responsive gene expression in skin after treatment with fresolimumab compared to pre-treatment TGF-beta responsive gene expression. | 7 weeks
  TGF-beta regulated skin gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lafyatis, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine; Rheumatology/Arthritis Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rice LM, Padilla CM, McLaughlin SR, Mathes A, Ziemek J, Goummih S, Nakerakanti S, York M, Farina G, Whitfield ML, Spiera RF, Christmann RB, Gordon JK, Weinberg J, Simms RW, Lafyatis R. Fresolimumab treatment decreases biomarkers and improves clinical symptoms in systemic sclerosis patients. J Clin Invest. 2015 Jul 1;125(7):2795-807. doi: 10.1172/JCI77958. Epub 2015 Jun 22. PMID 26098215